CLINICAL TRIAL: NCT03036072
Title: Delayed Rewarming for Neuroprotection in Infants Following Cardiopulmonary Bypass Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexa Craig (Other)
Collaborators: MaineHealth (Other)
Responsible Party: Sponsor-Investigator, Alexa Craig, Assistant Professor of Pediatrics, MaineHealth
Organization: MaineHealth (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB 4489; 4KL2TR001063-04 (NIH)
Record Dates: First submitted 2017-01-24; First posted 2017-01-30 (Estimated); Results first posted 2020-04-15 (Actual); Last update posted 2020-07-13 (Actual); Status verified 2020-04

CONDITIONS: Post-Op Complication
Keywords: Therapeutic Hypothermia
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Strict Normothermia (Active Comparator): Patients will be rewarmed to 36.5 degrees centigrade in the operating room and maintained here by conventional means in the PICU.
  Interventions: Other: Strict normothermia
- Delayed Rewarming (Experimental): Patient will be rewarmed to 35.0 degrees centigrade in the operating room, then slowly rewarmed to normal physiologic temperature over 12 hours by using a servo-controlled cooling blanket. Normothermia will be maintained by the cooling blanket for an additional 12 hours.
  Interventions: Device: Delayed Rewarming

INTERVENTIONS:
Other: Strict normothermia
  Arms: Strict Normothermia
Device: Delayed Rewarming — Use of the servo-controlled cooling blanket for delayed rewarming to target temperature.
  Arms: Delayed Rewarming

SUMMARY:
This is an unblinded, single center, randomized study of infants with congenital heart disease undergoing cardiopulmonary bypass surgery, randomized to either the delayed rewarming intervention or to the standard of care (strict normothermia).

DETAILED DESCRIPTION:
Control Group:

The congenital heart surgery will be performed according to usual practice with the degree of intra-operative hypothermia determined by the cardiothoracic surgeon based on the anticipated complexity of the case. Following completion of the surgical procedure, the infant will be rapidly rewarmed on CPB at a rate of 0.2 to 0.3°C per minute to a normothermic temperature of 36.5°C. Infants in this group will be given a single weight-based 15 mg/kg dose of intravenous Tylenol in the operating room (OR) by the anesthesiologist as the chest is being closed. The infant will be transported to the Pediatric Intensive Care Unit (PICU) for routine post-operative monitoring. If the infant develops a fever, ice packs will be applied to the axilla and groin per usual routine and removed once the fever has abated.

Experimental group:

Partial rewarming will occur on CPB to 35°C. During the last hour of surgery, the infant's temperature will be maintained at 35°C while the chest is closed by using a BairHugger and lowering the room temperature. Transfusions of packed red blood cells, fresh frozen plasma and cryoprecipitate will not be automatically warmed. Infants will be given a single 15 mg/kg dose of IV Tylenol in the OR. The infant will be transported to the PICU at 35°C and placed on the temperature-regulating blanket. The infant will be incrementally rewarmed with increases in temperature of 0.3°C every 2 hours for 6 hours, then 0.2°C every 2 hours for 6 hours to the goal temperature of 36.5°C. Once the infant is stable, EEG will be performed for 48 hours to screen for seizures. The PI will interpret the EEG every 6-8 hours. The infant will remain on the blanket at 36.5°C for another 12 hours. The blanket and esophageal temperature probe will then be removed a total of 24 hours after surgery was completed.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of congenital heart disease requiring congenital heart surgery on bypass
2. Age less than 6 months at the time of surgery
3. Intra-operative hypothermia less than or equal to 35°C

Exclusion Criteria:

1. Concern for underlying coagulation disorder such as hemophilia
2. Death in the operating room
3. Inability to wean of cardiopulmonary bypass at conclusion of surgery

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2019-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexa K Craig, MD, MSc, Principal Investigator — Assistant Professor of Pediatrics
Locations (1):
- Maine Medical Center, Portland, Maine, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Strict Normothermia: Patients will be rewarmed to 36.5 degrees centigrade in the operating room and maintained here by conventional means in the PICU.
  Strict normothermia
- Delayed Rewarming: Patient will be rewarmed to 35.0 degrees centigrade in the operating room, then slowly rewarmed to normal physiologic temperature (36.5) over 12 hours by using a servo-controlled cooling blanket. Normothermia will be maintained by the cooling blanket for an additional 12 hours.
  Delayed Rewarming: Use of the servo-controlled cooling blanket for delayed rewarming to target temperature.
Period: Overall Study
Arm/Group | Strict Normothermia | Delayed Rewarming
Started | 12 | 13
Completed | 12 | 10
Not Completed | 0 | 3
Not completed — Death | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Strict Normothermia | Delayed Rewarming | Total
Number analyzed (Participants) | 12 | 10 | 22
Age, Customized [Count of Participants; unit: Participants]
  Less than 2 weeks at surgery | 4 | 3 | 7
  More than 2 weeks at surgery | 8 | 7 | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 8 | 6 | 14
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 10 | 8 | 18
  Unknown | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 12 | 10 | 22
Trisomy 21 [Count of Participants; unit: Participants] | 4 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: Infants With Elevated s100b and NSE
Description: In a population of infants with congenital heart disease undergoing cardiopulmonary bypass surgery, does delayed rewarming administered during the 12 hours after surgery, compared to standard care, decrease brain injury as measured by levels of serum biomarkers of brain injury, s100b and neuron specific enolase during the four days after surgery?
Time Frame: 4 days
Population: Laboratory storage and transportation issues resulted in less than expected number of viable specimens that could be analyzed at all 5 time points.
Measure: Count of Participants; unit: Participants
Arm/Group | Strict Normothermia | Delayed Rewarming
Number analyzed (Participants) | 12 | 10
Participants | 11 | 9

2. Secondary Outcome: Number of Participants With Adverse Events
Description: In a population of infants with congenital heart disease undergoing cardiopulmonary bypass surgery, is there evidence for increased frequency of severe, moderate or other adverse events in the delayed rewarming group compared to the standard of care group?
Time Frame: 4 days
Measure: Count of Participants; unit: Participants
Arm/Group | Strict Normothermia | Delayed Rewarming
Number analyzed (Participants) | 12 | 10
Participants | 3 | 3

ADVERSE EVENTS:
Time Frame: Until 48 hours post surgery.
Arm/Group | Strict Normothermia | Delayed Rewarming
All-Cause Mortality (participants affected / at risk) | 0/12 | 1/10
Serious Adverse Events (participants affected / at risk) | 3/12 | 2/10
Other Adverse Events (participants affected / at risk) | 0/12 | 0/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Strict Normothermia (N=12) | Delayed Rewarming (N=10)
ECMO after surgery (Cardiac disorders) | 1 (1) | 1 (1) — Patient unable to wean from bypass following surgery.
CPR after surgery (Cardiac disorders) | 1 (1) | 0 (0)
Return to Operating Room (Cardiac disorders) | 3 (3) | 1 (1)
Stroke or Seizure (Nervous system disorders) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-31): https://cdn.clinicaltrials.gov/large-docs/72/NCT03036072/Prot_SAP_000.pdf